CLINICAL TRIAL: NCT01676571
Title: A Single-centre, Open-label, Single-dose Interventional Study Investigating the Pharmacokinetic Properties of Lu AA21004 in Healthy Young Chinese Men and Women
Brief Title: Pharmacokinetic Properties of Lu AA21004 (Vortioxetine) in Healthy Young Chinese Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14077A
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lu AA21004 (Experimental)
  Interventions: Drug: Lu AA21004

INTERVENTIONS:
Drug: Lu AA21004 — 10 mg immediate-release (IR), one single dose, orally
  Other Names: Vortioxetine

SUMMARY:
The rationale for this pharmacokinetic (PK) study is to determine the PK parameters for Lu AA21004 (Vortioxetine) in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a Chinese man or woman
* The subject is, in the opinion of the investigator, generally healthy
* If female, the subject must have a negative pregnancy test at screening and baseline, and agree not to try to become pregnant from Screening until after the Follow-up Visit

Exclusion Criteria:

* The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
PK AUC determination of Lu AA21004 (Vortioxetine) | 11 days
  Area under the curve (AUC)
PK Cmax determination of Lu AA21004 (Vortioxetine) | 11 days
  Maximum observed concentration (Cmax)

OTHER OUTCOMES:
PK MR determination of metabolites Lu AA34443 and Lu AA39835 | 11 days
  Metabolic ratio (MR)
Number of patients with adverse events as a measure of safety and tolerability | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- CN001, Tianjin, China

REFERENCES:
- [Derived] Miao J, Wang G, Hou J, Areberg J, Zhao Y, Hojer AM, Ettrup A. Pharmacokinetics and Safety of Vortioxetine in the Chinese Population. Adv Ther. 2019 Nov;36(11):3134-3146. doi: 10.1007/s12325-019-01092-4. Epub 2019 Sep 24. PMID 31552551